CLINICAL TRIAL: NCT03684265
Title: An Open-label, Randomised, Single-dose, Two-way Crossover Study in Healthy Male and Female Volunteers to Evaluate the Relative Bioavailability of a New Oral Formulation of Meloxicam, Movalis® Capsules 15 mg, Versus Movalis® Tablets 15 mg, After Administration Under Fasting State.
Brief Title: A Study to Compare the Amount of Meloxicam in the Blood When it is Taken as Capsules or as Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0107-0277
Record Dates: First submitted 2018-09-24; First posted 2018-09-25 (Actual); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Healthy
MeSH Terms: interventions — Meloxicam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test to Reference (Experimental)
  Interventions: Drug: Meloxicam Capsule (Test); Drug: Meloxicam Tablet (Reference)
- Reference to Test (Experimental)
  Interventions: Drug: Meloxicam Capsule (Test); Drug: Meloxicam Tablet (Reference)

INTERVENTIONS:
Drug: Meloxicam Capsule (Test) — single dose
  Other Names: Movalis
Drug: Meloxicam Tablet (Reference) — single dose
  Other Names: Movalis

SUMMARY:
The primary objective of the study is to investigate the relative bioavailability of Movalis capsules 15 mg (Test, T) versus Movalis tablets 15 mg (Reference, R).

The secondary objective of the study is to establish bioequivalence of Movalis capsules 15 mg (Test, T) versus Movalis tablets 15 mg (Reference, R).

ELIGIBILITY:
Inclusion criteria:

* Male and female subjects aged 18-45, inclusive.
* Body mass index by Quetelet between 18.50 -29.99 kg/m2, inclusive.
* The verified diagnosis is "healthy" according to the conclusion investigator according to the information in the anamnesis, the results of the physical examination, the Electrocardiogram (ECG), the results of measurement of vital signs of the body (blood pressure, heart rate, breathing rate and body temperature), and laboratory indicators.
* Pre-conducting standard clinical and laboratory and instrumental studies did not reveal the presence of any diseases and abnormalities.
* Systolic blood pressure not less than 100 mm Hg. and not higher than 139 mm Hg. diastolic blood pressure not less than 70 mm Hg. and not more than 90 mm Hg. the heart rate is not less than 60 beats per minute and not more than 90 beats per minute, the frequency of respiratory movements is within the range of 12-20 per minute.
* Ability to understand and accept the explanation of the study; the written informed consent of the volunteer to participate in the study in accordance with applicable law.
* Female subjects of childbearing potential who agree on using double-barrier contraception from a screening visit to 30 days after the last administration of the study drug, inclusive. If a female is postmenopausal (no menses for at least 1 year) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) she will be exempt from the requirement. In case of using oral contraceptives, these should be withdrawn at least 2 months before the study.
* Male subjects who agree on using effective contraception (barrier contraceptive methods) from a screening visit to 30 days after the last administration of the study drug, inclusive.

Exclusion criteria:

* Drug intolerance of any drug.
* Allergic history.
* Acute infectious diseases or allergic reactions requiring treatment (including drug allergy), less than 4 weeks before the screening.
* Surgical interventions on the gastrointestinal tract (with the exception of appendectomy), which can have a significant effect on the absorption or metabolism of study drugs.
* Known hypersensitivity to meloxicam or any excipient of the test and reference products.
* Known hypersensitivity to other Non-steroid anti-inflammatory drug (NSAIDs): subjects who have developed signs of asthma, nasal polyps, angio-oedema or urticarial following the administration of acetylsalicylic acid or other NSAIDs.
* Chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine system, as well as diseases of the gastrointestinal tract, liver, kidneys, blood, or other conditions that make it impossible for the volunteer to participate in the study according to the investigator opinion.
* The results of standard laboratory and instrumental methods of examination, obtained during the screening, go beyond normal values.
* History of gastro-intestinal ulceration/ perforation or bleeding; history of malignancy within 5 years before the screening.
* Positive results of blood tests for infections (HIV, syphilis, hepatitis B or C) at screening.
* A positive alcohol test at screening.
* A positive urine drug test (cannabis, benzodiazepines, barbiturates, opiates, cocaine, and amphetamines) at screening.
* Pregnancy or breastfeeding.
* Any diet, for example, vegetarian, for 2 weeks before the first day of screening.
* Alcohol intake more than 10 units. alcohol per week (1 unit of alcohol is equivalent to ½ liter of beer, 200 ml of wine or 50 ml of alcohol) or anamnestic information about alcoholism, drug addiction, abuse of medicines.
* The inability to be without food for at least 12 hours and the inability to take the drug on an empty stomach.
* Blood donation (≥ 450 ml) within 3 months before screening.
* Depot injections, the installation of intrauterine hormonal therapy systems or implants of any drugs for 6 months before the screening;
* For women: use of hormonal contraceptives less than 2 months before the screening.
* Regular drug intake within 2 weeks before the screening.
* Intake of systemic drugs known to alter liver function (barbiturates, omeprazole, cimetidine) within 4 weeks before the screening.
* For women: volunteers with preserved reproductive potential who had unprotected intercourse with an unsterilized male partner for 30 days before the screening
* Participation in another clinical trial within 3 months before the screening.
* Difficult access to the vein, complicating or making it impossible to install a catheter and frequent blood sampling.
* Smoker (≥10 cigarettes or ≥ 3 pipes per day).
* Inability to refrain from smoking on study days.
* Volunteers who do not want or are unable to give up alcohol and excessive physical exertion from the first day of screening and before the visit of follow-up.
* Volunteers who are unwilling or unable to refuse drinks and food containing methylxanthines (coffee, tea, cola, energy drinks, chocolate, etc.) and grapefruit / grapefruit juice, Seville oranges (sour or bitter oranges) and their juices, and dietary supplements and products including St. John's wort (Hypericum perforatum) from the first day of screening and until a follow-up visit.
* Volunteers who lead a lifestyle (including night work and extreme physical activities such as sports or weight lifting), which can make it difficult to interpret the laboratory data obtained during the study.
* Volunteers who do not intend to comply with the study regime.
* Volunteers who are obviously or probably, in the opinion of the investigator, are not able to understand and evaluate the information on this study in the process of signing the ICF, in particular regarding the expected risks and possible discomfort.
* The presence of volunteers dehydration due to diarrhea, vomiting or other cause within the last 24 hours before the first day of screening.
* The presence of volunteers attacks of seizures, epilepsy and any other neurological disorders in the anamnesis
* Recent cerebrovascular bleeding or established systemic bleeding disorders.
* Known lactose intolerance.
* Reports difficulty for swallowing tablets or capsules.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- City Clinical Hospital named after V.P. Demikhova Department of Health of Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). Requestors can use the following link http:// trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement'.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was a randomised, two-period, two sequences, single-dose, open-label, and crossover trial in healthy male and female subjects in fasting conditions.
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist site to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial drug if any of the specific entry criteria was violated. In this study, 26 subjects were entered & treated.
Groups:
- Movalis® Capsules (T), Then Movalis® Tablets (R): Patient were orally administered single dose of Movalis® capsules 15 mg (T) with 200 mL of water after an overnight fast of at least 10 hours (h) in Period 1, followed with single dose of Movalis® tablets 15 mg (R) with 200 mL of water after an overnight fast of at least 10 h in Period 2.
  The washout period between two drug administrations was of 7 days.
- Movalis® Tablets (R), Then Movalis® Capsules (T): Patient were orally administered single dose of Movalis® tablets 15 mg (R) with 200 mL of water after an overnight fast of at least 10 h in Period 1, followed with single dose of Movalis® capsules 15 mg (T) with 200 mL of water after an overnight fast of at least 10 h in Period 2.
  The washout period between two drug administrations was of 7 days.
Period: Treatment Period 1
Arm/Group | Movalis® Capsules (T), Then Movalis® Tablets (R) | Movalis® Tablets (R), Then Movalis® Capsules (T)
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Washout Period of 1 Week
Arm/Group | Movalis® Capsules (T), Then Movalis® Tablets (R) | Movalis® Tablets (R), Then Movalis® Capsules (T)
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Movalis® Capsules (T), Then Movalis® Tablets (R) | Movalis® Tablets (R), Then Movalis® Capsules (T)
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Movalis® Capsules (T), Then Movalis® Tablets (R) | Movalis® Tablets (R), Then Movalis® Capsules (T) | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.5 (7.4) | 29.5 (6.0) | 30.0 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 3 | 2 | 5
Race/Ethnicity, Customized [Number; unit: Paticipants] — All subjects were Caucasian. Ethnicity were not collected from any participant
  Paticipants
    Caucasian | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-t)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-t).
  Standard error is actually Geometric standard error.
Time Frame: Baseline (pre-dose), 0.5 hours (h), 1.0h, 2.0h, 3.0h, 4.0h, 5.0h, 6.0h, 7.0h, 8.0h, 10.0h, 12.0h, 24.0h, 32.0h, 48.0h and 72.0h post-dose
Population: Pharmacokinetic set (PKS): This set includes all randomised subjects who met the protocol requirements without important protocol deviation and completed all study periods.
Measure: Geometric Least Squares Mean (Standard Error); unit: Nanogram (ng)·hour (h)/ mililiter(mL)
Groups:
- Movalis® Capsules (T): Patient were orally administered single dose of Movalis® capsules 15 mg (T) with 200 mL of water after an overnight fast of at least 10 h.
- Movalis® Tablets (R): Patient were orally administered single dose of Movalis® tablets 15 mg (R) with 200 mL of water after an overnight fast of at least 10 h.
Arm/Group | Movalis® Capsules (T) | Movalis® Tablets (R)
Number analyzed (Participants) | 26 | 26
Nanogram (ng)·hour (h)/ mililiter(mL) | 27870.56 (1.06) | 30051.25 (1.06)
Statistical Analysis 1: Comparison: Movalis® Capsules (T) vs Movalis® Tablets (R); Relative bioavailability comparison of Movalis® capsules (T) with Movalis® tablets (R) for AUC0-t. The analysis of variance (ANOVA) model in the log scale was used. This model included the sequence, period and type of therapy as fixed effects and the effect study subjects grouped within the sequence was considered random; Test type: Equivalence — Bioequivalence acceptance range for the ratio of geometric means was 80- 125%; Geometric mean ratio T/R, % = 92.74, 95% CI 2-sided [89.02 to 96.62], Standard Error of Mean 8.66 — Standard error of the mean is actually intra individual coefficient of variation

2. Primary Outcome: Maximum Measured Concentration of the Analyte in Plasma (Cmax)
Description: Maximum measured concentration of the analyte in plasma (Cmax).
  Standard error is actually Geometric standard error.
Time Frame: Baseline (pre-dose), 0.5 hours(h), 1.0h, 2.0h, 3.0h, 4.0h, 5.0h, 6.0h, 7.0h, 8.0h, 10.0h, 12.0h, 24.0h, 32.0h, 48.0h and 72.0h post-dose
Population: PKS
Measure: Geometric Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Movalis® Capsules (T) | Movalis® Tablets (R)
Number analyzed (Participants) | 26 | 26
ng/mL | 1131.12 (1.04) | 1432.83 (1.04)
Statistical Analysis 1: Comparison: Movalis® Capsules (T) vs Movalis® Tablets (R); Relative bioavailability comparison of Movalis® capsules (T) with Movalis® tablets (R) for Cmax. The analysis of variance (ANOVA) model in the log scale was used. This model included the sequence, period and type of therapy as fixed effects and the effect study subjects grouped within the sequence was considered random; Test type: Equivalence — Bioequivalence acceptance range for the ratio of geometric means was 80- 125%; Geometric mean ratio T/R, % = 78.94, 90% CI 2-sided [73.70 to 84.56], Standard Error of Mean 14.57 — Standard error of the mean is actually intra individual coefficient of variation

3. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  Standard error is actually Geometric standard error.
Time Frame: as for outcome 2
Population: PKS
Measure: Geometric Least Squares Mean (Standard Error); unit: ng·h/mL
Arm/Group | Movalis® Capsules (T) | Movalis® Tablets (R)
Number analyzed (Participants) | 26 | 26
ng·h/mL | 32863.87 (1.09) | 33867.43 (1.09)
Statistical Analysis 1: Comparison: Movalis® Capsules (T) vs Movalis® Tablets (R); Relative bioavailability comparison of Movalis® capsules (T) with Movalis® tablets (R) for AUC0-∞. The analysis of variance (ANOVA) model in the log scale was used. This model included the sequence, period and type of therapy as fixed effects and the effect study subjects grouped within the sequence was considered random; Test type: Equivalence — Bioequivalence acceptance range for the ratio of geometric means was 80- 125%; Geometric mean ratio T/R, % = 97.04, 90% CI 2-sided [92.57 to 101.72], Standard Error of Mean 9.96 — Standard error of the mean is actually intra individual coefficient of variation

ADVERSE EVENTS:
Time Frame: From first drug administration until 7 days after the last drug administration, ie., up to 8 days.
Description: There were no Serious Adverse Event (SAE), Death and other Adverse Event (AE) (with frequency threshold of 5%) were reported for this tiral.
Arm/Group | Movalis® Capsules (T) | Movalis® Tablets (R)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT03684265/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT03684265/SAP_001.pdf